CLINICAL TRIAL: NCT00092482
Title: Immunogenicity and Safety of Gardasil (V501) Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Consistency Lots for 16- to 23-Year-Old Women With and Additional Immunogenicity Bridge to the Monovalent HPV 16 Vaccine Pilot Manufacturing Lot Study-The F.U.T.U.R.E. Study (Females United to Unilaterally Reduce Endo/Ectocervical Disease)
Brief Title: Immunogenicity Bridge Between an Investigational Monovalent Vaccine and the Equivalent Component of Gardasil (V501) a Quadrivalent Vaccine (V501-012)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-012; 2004_080
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cervical Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine / Duration of Treatment: 4 years

SUMMARY:
The purpose of the study is to determine if an investigational vaccine with a single component develops an immune response that is similar to the equivalent investigational vaccine with four components to reduce cervical disease.

ELIGIBILITY:
Inclusion Criteria:

* Female with an intact uterus with lifetime history of 0-4 sexual partners

Exclusion Criteria:

* Prior Human Papillomavirus Vaccine (HPV) vaccination;
* Prior abnormal paps;
* Prior history of genital warts

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3882 (Actual)
Dates: Start 2002-06-28 (Actual); Primary Completion 2004-06-30 (Actual); Study Completion 2008-08-15 (Actual)

PRIMARY OUTCOMES:
Tolerability and immune responses at week 4 post dose 3.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Garland SM, Steben M, Hernandez-Avila M, Koutsky LA, Wheeler CM, Perez G, Harper DM, Leodolter S, Tang GW, Ferris DG, Esser MT, Vuocolo SC, Nelson M, Railkar R, Sattler C, Barr E; 012 Study Investigators. Noninferiority of antibody response to human papillomavirus type 16 in subjects vaccinated with monovalent and quadrivalent L1 virus-like particle vaccines. Clin Vaccine Immunol. 2007 Jun;14(6):792-5. doi: 10.1128/CVI.00478-06. Epub 2007 Apr 11. PMID 17428949
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- [Result] Brown DR, Garland SM, Ferris DG, Joura E, Steben M, James M, Radley D, Vuocolo S, Garner EI, Haupt RM, Bryan JT. The humoral response to Gardasil over four years as defined by total IgG and competitive Luminex immunoassay. Hum Vaccin. 2011 Feb;7(2):230-8. doi: 10.4161/hv.7.2.13948. Epub 2011 Feb 1. PMID 21307649
- [Derived] Brown DR, Castellsague X, Ferris D, Garland SM, Huh W, Steben M, Wheeler CM, Saah A, Luxembourg A, Li S, Velicer C. Human papillomavirus seroprevalence and seroconversion following baseline detection of nine human papillomavirus types in young women. Tumour Virus Res. 2022 Jun;13:200236. doi: 10.1016/j.tvr.2022.200236. Epub 2022 May 4. PMID 35525430
- [Derived] Doshi P, Bourgeois F, Hong K, Jones M, Lee H, Shamseer L, Spence O, Jefferson T. Adjuvant-containing control arms in pivotal quadrivalent human papillomavirus vaccine trials: restoration of previously unpublished methodology. BMJ Evid Based Med. 2020 Dec;25(6):213-219. doi: 10.1136/bmjebm-2019-111331. Epub 2020 Mar 17. PMID 32184277
- [Derived] Insinga RP, Perez G, Wheeler CM, Koutsky LA, Garland SM, Leodolter S, Joura EA, Ferris DG, Steben M, Hernandez-Avila M, Brown DR, Elbasha E, Munoz N, Paavonen J, Haupt RM; FUTURE I Investigators. Incident cervical HPV infections in young women: transition probabilities for CIN and infection clearance. Cancer Epidemiol Biomarkers Prev. 2011 Feb;20(2):287-96. doi: 10.1158/1055-9965.EPI-10-0791. PMID 21300618
- [Derived] Garland SM, Insinga RP, Sings HL, Haupt RM, Joura EA. Human papillomavirus infections and vulvar disease development. Cancer Epidemiol Biomarkers Prev. 2009 Jun;18(6):1777-84. doi: 10.1158/1055-9965.EPI-09-0067. PMID 19505910
- [Derived] Brown DR, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, Sings HL, James M, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in generally HPV-naive women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):926-35. doi: 10.1086/597307. PMID 19236279
- [Derived] Wheeler CM, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, James M, Vuocolo S, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in sexually active women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):936-44. doi: 10.1086/597309. PMID 19236277
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html